CLINICAL TRIAL: NCT05615935
Title: The Effects of Experiential HIV Testing to Improve Knowledge and Practice, and Reduce Stigma Toward HIV of Emergency Department Nurses
Brief Title: Experiential HIV Testing Increasing Testing Related Knowledge and Practice, and Reduce Stigma Toward HIV of Nurses.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University (Other)
Responsible Party: Principal Investigator, Piao-Yi Chiou, Associate Professor, National Taiwan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 202209065RINA
Record Dates: First submitted 2022-10-31; First posted 2022-11-14 (Actual); Results first posted 2024-08-02 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Hiv; HIV Testing
Keywords: stigma; knowledge; Education, nursing; situated learning
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Social Stigma

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Get a learning material and a experiential HIV Testing (Experimental): These participants in the experimental group will be provided a learning material about HIV testing, then an experiential HIV Testing, which includes HIV testing and counselling, education and discussion, and a post-test interviews will be provided.
  Interventions: Other: Experiential HIV Testing
- Get a learning material only (No Intervention): These participants in the control group will be provided a learning material about HIV testing only. After the post-test, the experiential HIV Testing will be provided to them.

INTERVENTIONS:
Other: Experiential HIV Testing — The content of experiential HIV Testing includes HIV testing, counselling, and education and discussion.
  Arms: Get a learning material and a experiential HIV Testing

SUMMARY:
This is a randomized controlled trial design. The investigators plan to recruit about 60 to 70 emergency department nurses from a medical center in Taipei, Taiwan. After completing the paper consent form, these nurses will be randomly assigned to 2 groups, which are a control group and an experimental group. The pre-test includes the demographic data sheet, HIV testing related knowledge and practice scale, and The Health Care Provider HIV/ AIDS Stigma Scale (HPASS). All nurses will receive a learning material when they finish the pre-test. In addition, the experimental group will be provided a real HIV testing and counselling by a researcher. The post-test will be finished one month later of pre-test in the control group, and one month later while the intervention completed in the experimental group. The semi-structural interview will be performed to the experimental group to collect and analyze their opinion toward the experiential HIV testing.

DETAILED DESCRIPTION:
This project aims to develop an intervention of "experiential HIV testing" and to verify the following effects on emergency nurses: (1) Improve HIV testing related knowledge and practice; (2) Reduce HIV-related stigma; (3) Find out the possible demographic factors that might affect the effectiveness of experiential HIV Testing. During the intervention, nurses can directly participate in the whole process of anonymous HIV testing in the role of who need to be screened, and pre- and post-testing counselling accompanied the education and discussion will also be provided to them by a researcher. Through the above-mentioned measures, the knowledge and practices related to the HIV testing could be improved, and the stigma attitude toward HIV could be reduced through the self-reflection on the testing process.

ELIGIBILITY:
Inclusion Criteria:

- have registered nurse license and do clinical care in emergency department

Exclusion Criteria:

* have registered nurse license but doesn't do clinical care, likes head nurse.
* do clinical care in emergency department but doesn't have registered nurse license, like volunteers or assistant nurse.
* have experienced non-occupational HIV testing.
* had been a nurse in HIV/AIDS-focus ward or HIV/AIDS case manager.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2022-11-09 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: CHENG-RU HE, Bachelor, Principal Investigator — National Taiwan University Hospital
Locations (1):
- School of Nursing of National Taiwan University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] He CR, Chang JC, Liu CY, Yang BJ, Hung YH, Chiou PY. Enhancing HIV knowledge and reducing stigma among emergency nurses through experiential self-testing: A mixed-methods study. Nurse Educ Pract. 2025 Dec 18;91:104694. doi: 10.1016/j.nepr.2025.104694. Online ahead of print. PMID 41455361

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Get a Learning Material and a Experiential HIV Testing | Get a Learning Material Only
Started | 37 | 37
Completed | 36 (on a long vacation) | 36 (lost contact (the participant didn't reply any message))
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Get a Learning Material and a Experiential HIV Testing | Get a Learning Material Only | Total
Number analyzed (Participants) | 36 | 36 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.03 (4.58) | 29.14 (5.74) | 28.58 (5.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 28 | 56
  Male | 8 | 8 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 36 | 36 | 72
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Taiwan | 36 | 36 | 72
education level [Count of Participants; unit: Participants]
  bachelor's degree | 33 | 33 | 66
  master's degree | 3 | 3 | 6
Marital status [Count of Participants; unit: Participants]
  married | 4 | 6 | 10
  single | 32 | 30 | 62
Nursing practice years [Mean (Standard Deviation); unit: years] | 5.06 (4.49) | 6.18 (5.28) | 5.62 (4.90)
Nursing practice years in the ED [Mean (Standard Deviation); unit: years] | 3.6 (3.64) | 4.77 (4.32) | 4.18 (4.01)
religion [Count of Participants; unit: Participants]
  Buddhism | 3 | 7 | 10
  Taoism | 6 | 6 | 12
  Buddhism and Taoism | 1 | 2 | 3
  Christianity | 2 | 2 | 4
  Catholicism | 1 | 0 | 1
  None | 23 | 19 | 42
catastrophic illness [Count of Participants; unit: Participants] — An acute or prolonged illness usually considered to be life-threatening or with the threat of serious residual disability
  Participants
    yes | 0 | 1 | 1
    no | 36 | 35 | 71
receiving HIV-related lecture in recent 12 months [Count of Participants; unit: Participants]
  yes | 11 | 10 | 21
  no | 25 | 26 | 51
ever had HIV occupational exposure or not [Count of Participants; unit: Participants]
  yes | 11 | 11 | 22
  no | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: HIV Testing Related Knowledge and Practice
Description: A self-development scale, known as the "HIV Testing-Related Knowledge and Practice Scale," is employed to assess individuals' knowledge and practices pertaining to HIV testing. The scale consists of twenty-eight questions, encompassing both True-False and multiple-choice formats. Participants earn one point for each correct answer, contributing to a total score that ranges from the minimum scores of 0 to the maximum scores of 28. Higher scores signify a more positive outcome, indicating enhanced HIV testing-related knowledge and practice among the participants.
Time Frame: pre-test(Baseline) and post-test (week 4)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Get a Learning Material and a Experiential HIV Testing | Get a Learning Material Only
Number analyzed (Participants) | 36 | 36
score on a scale
  pre-test | 17.17 (1.88) | 17.22 (2.14)
  post-test | 19.44 (2.21) | 17.36 (2.69)
Statistical Analysis 1: Comparison: Get a Learning Material and a Experiential HIV Testing vs Get a Learning Material Only; Using G*Power 3.1, the required sample size for ANCOVA with two groups was estimated with a significance level of 0.05, statistical power of 0.80, and an effect size of 0.35, based on Cohen's guidelines for a medium-to-large effect commonly applied in behavioral research (Cohen, 1988). Assuming up to two covariates, a minimum of 67 participants was required. Accounting for a 10% attrition rate, the final target was set at 74 participants; Test type: Superiority; p < 0.001, ANCOVA — The p-value is adjusted for multiple comparisons using the Bonferroni correction, with a significance threshold of 0.05; Adjusted Mean Difference (ANCOVA) = 2.07

2. Primary Outcome: HIV Related Stigma
Description: The Healthcare Provider HIV/AIDS Stigma Scale (HPASS) will be used to assess this outcome. The instrument contains 30 items, each scored on a six-point Likert scale, yielding a minimum total score of 30 and a maximum of 180. Higher scores reflect greater levels of stigma toward people living with HIV, indicating a worse outcome. Validation of the HPASS through factor analysis identified three underlying dimensions. The stereotyping dimension (11 items; score range: 11-66) reflects negative cognitions and beliefs about people living with HIV. The prejudice dimension (13 items; score range: 13-78) captures emotionally driven attitudes. The discrimination dimension (6 items; score range: 6-36) represents behavioral responses stemming from negative attitudes. For all dimensions, higher scores indicate worse outcomes. These 3 dimensions(as sub-scale scores) for stereotyping, prejudice, and discrimination will also be calculated and analyzed.
Time Frame: pre-test (Baseline) and post-test (Week 4)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Get a Learning Material and a Experiential HIV Testing | Get a Learning Material Only
Number analyzed (Participants) | 36 | 36
score on a scale
  (pre-test)HPASS in total | 89.39 (16.14) | 86.75 (22.06)
  (post-test)HPASS in total | 85.94 (20.10) | 88.03 (20.44)
  (pre-test)stereotyping | 36.36 (6.85) | 38.36 (8.43)
  (post-test)stereotyping | 36.31 (7.66) | 38.03 (9.20)
  (pre-test)prejudice | 35.78 (8.51) | 34.44 (12.11)
  (post-test)prejudice | 33.14 (10.73) | 34.72 (10.31)
  (pre-test)discrimination | 17.25 (5.61) | 13.94 (5.68)
  (post-test)discrimination | 16.50 (5.59) | 15.28 (5.32)
Statistical Analysis 1: Comparison: Get a Learning Material and a Experiential HIV Testing vs Get a Learning Material Only; Test type: Superiority; p = 0.15, ANCOVA — The p-value is adjusted for multiple comparisons using the Bonferroni correction, with a significance threshold of 0.05; Adjusted Mean Difference (ANCOVA) = 4.58
Statistical Analysis 2: Comparison: Get a Learning Material and a Experiential HIV Testing; Test type: Superiority; p = 0.02, t-test, 2 sided — The p-value is adjusted for multiple comparisons using the Bonferroni correction, with a significance threshold of 0.05; Median Difference (Final Values) = -2.64, Standard Deviation 6.35

ADVERSE EVENTS:
Time Frame: 1 year
Description: Due to the cross-sectional non-interventional nature of this study, participants will not be at risk for Serious Adverse Events, at risk for All-Cause Mortality, and at risk for Other (Not Including Serious) Adverse Events.
Arm/Group | Get a Learning Material and a Experiential HIV Testing | Get a Learning Material Only
All-Cause Mortality (participants affected / at risk) | 0/72 | 0/72
Serious Adverse Events (participants affected / at risk) | 0/72 | 0/72
Other Adverse Events (participants affected / at risk) | 0/72 | 0/72

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-20): https://cdn.clinicaltrials.gov/large-docs/35/NCT05615935/Prot_SAP_000.pdf